CLINICAL TRIAL: NCT03377946
Title: Effect of Probiotics on Pre-diabetes and Diabetes in China-the Role of Gut Microbiota Composition
Brief Title: Effect of Probiotics on Pre-diabetes and Diabetes in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zeng, Director of Health Management Institue, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHPF2017019
Record Dates: First submitted 2017-12-10; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: pre-diabetes,diabetes,probiotics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- probiotics on type 2 diabetes (Experimental): take probiotics
  Interventions: Biological: probiotics
- probiotics on pre-diabetes (Experimental): take probiotics
  Interventions: Biological: probiotics
- placebo on type 2 diabetes (Placebo Comparator): take placebo
  Interventions: Biological: placebo
- placebo on pre-diabetes (Placebo Comparator): take placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: probiotics — the probiotics group was taking probiotics 4 packets a day
  Arms: probiotics on pre-diabetes; probiotics on type 2 diabetes
Biological: placebo — the placebo group was taking placebo 4 packets a day
  Arms: placebo on pre-diabetes; placebo on type 2 diabetes

SUMMARY:
This study is aimed at verifying the effects of probiotics (KAWAI:dead S.thermophilus) on glucos management among T2DM and pre-diabetes Chinese adult. Additionally, the investigators intend to verify the effects of probiotics on modifying the structure and function of gut microbiome.

DETAILED DESCRIPTION:
Methods: double-blind, randomized controlled trial. Number of participants: 160 patients with pre-diabetes and 60 diabetes. Intervention time: 3months. Data and Specimen collection time: at baseline and after the intervention.

Observation index

1. Physical measurement: gender, age, weight, BMI, waist circumference, hip circumference, waist-to-hip ratio, systolic pressure, diastolic blood pressure.
2. Lifestyle questionnaire: diet, drinking, exercise, sleep and other habits.
3. Blood test: blood glucose, OGTT, blood lipid, TNF-a, il-6, il-10, LPS, glp-1, gut microbiome metabolism products, T2DM related methylation.

4. Gut microbiome detection: gut microbiome 16Sr DNA sequencing, gut microbiome bioinformatics analysis

ELIGIBILITY:
Inclusion Criteria:

1. Meet Diabetes/pre-diabetes diagnostic criteria
2. BMI 18-35kg/m2

Exclusion Criteria:

1. Patients with diabetes or hyperlipidemia, and need regular use of drugs.
2. Secondary obesity or diabetes
3. Digestive, tumor, heart, lung, kidney, rheumatic immunity and other systemic serious diseases
4. Pregnant women, women ready for pregnancy, and nursing mothers
5. Take antibiotics or bacterial agents within 1 month
6. Diarrhea or abscess in 1 month or blood or other abnormal feces
7. Diabetics have a history of more than 2 years
8. The OGTT experiment of diabetic patients FG≥9mmol/L or 2h≥14mmol/L

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-12-21 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes of blood glucose and insulin sensitivity | 3~5 years
  blood glucose of fasting and 2 hours after OGTT，fasting insulin
Changes of gut microbiota composition | 3~5 years
  Feces gut microbiome 16Sr DNA sequencing, gut microbiome bioinformatics analysis

SECONDARY OUTCOMES:
Changes of blood inflammatory markers | 3~5 years
  blood TNF-a, Il-6, Il-10, LPS
Composite changes in diabetes risk factors | 3~5 years
  blood pressure, triglyceride,Cholesterol,LDL,HDL, weight
Composite changes of weight, waist circumference and BMI | 3~5 years
  weight, waist circumference,BMI,body fat

OTHER OUTCOMES:
Changes of Intestinal endocrine function | 3~5 years
  Blood GLP-1

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zeng, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- health management center,Southwest hospital, Chongqing, Chongqing Municipality, China

DOCUMENTS (2):
  • Study Protocol (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03377946/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03377946/SAP_001.pdf